CLINICAL TRIAL: NCT06519006
Title: Effectiveness of Pelvic Floor Exercise to Prevent LARS (Low Anterior Resection Syndrome) After Mini-invasive Low Anterior Resection in Patients With Rectal Cancer
Brief Title: Effectiveness of Pelvic Floor Exercise to Prevent LARS (Low Anterior Resection Syndrome)
Acronym: CH1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: F. D. Roosevelt University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHIRURGIA2024
Record Dates: First submitted 2024-06-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Prevention; LARS - Low Anterior Resection Syndrome; Pelvic Floor Disorders; Rectal Cancer; Low Anterior Resection
Keywords: prevention, LARS, pelvic floor exercise, LAR
MeSH Terms: conditions — Low Anterior Resection Syndrome; Pelvic Floor Disorders; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group - usual management (No Intervention): This arm will be managed as usual - without specific pelvic floor exercises after surgery, and 1, 6 and 12 months after low anterior resection, patients will be questioned about the possible development of LARS.
- Intervention group - specific pelvic floor exercise after LAR (Experimental): This arm will be instructed to exercise pelvic floor after low anterior resection for one month and 1, 6, and 12 months postoperatively will be questioned about the possible development of LARS.
  One month after surgery they will also be questioned about adherence to prescribed exercise.
  Interventions: Procedure: Pelvic floor exercise

INTERVENTIONS:
Procedure: Pelvic floor exercise — Exercises aimed at this issue consist of identification and isolated contraction of the pelvic floor muscles as well as their activation during complex movements and daily activities. During the engagement of the pelvic floor muscles, the correct engagement of the respiratory activity is important. Within the exercise units, exercises are used from sphincter contraction, through the gradual activation of individual pelvic floor layers in various ways, to their complex involvement in movement activities. Exercises are practiced repeatedly, at different frequencies and intensities that gradually increase, 4-5 times per day.
  Arms: Intervention group - specific pelvic floor exercise after LAR

SUMMARY:
The main aim of this randomized study will be to determine the effectiveness of pelvic floor exercises on the incidence or severity of LAR syndrome in patients after mini-invasive rectal resection.

The main questions it aims to answer are:

* Does pelvic floor exercise after low anterior resection prevent LARS (low anterior resection syndrome)?
* What is the adherence of patients to prescribed home exercise after surgery?
* Quality of life after LAR

Researchers will compare the group of patients with pelvic floor exercises to those without and determine the occurrence and severity of LARS.

Participants will:

* under the professional guidance of a physiotherapist, the day before surgery and in the first 4 postoperative days be educated to exercise the pelvic floor
* continue exercise at home for a month (according to the instructions together with the infographic)

DETAILED DESCRIPTION:
Advances in the surgical treatment of rectal diseases lead to better oncological results, a higher chance of preserving the sphincters, and thus a lower number of permanent stomas. However, the preserved anus does not always have to perform its original function fully. All patients after a low anterior resection of the rectum are at risk of developing functional disorders, the so-called LARS (low anterior resection syndrome). Patients may develop varying degrees of functional anorectal disorder, from urgency, stool incontinence to constipation. The prevalence of LARS ranges from 41-80% and is a significant factor in reducing the quality of life.

The therapy of LAR syndrome, depending on the severity, consists of medication, transanal irrigation, pelvic floor rehabilitation, neurostimulation or surgery. The most effective is a combination of treatment modalities. Given the lack of high-quality evidence in this area, recommendations are generally based on retrospective studies or extrapolated from studies of non-surgical patients with similar gastrointestinal disorders. Suppose the disease is present 1-2 years after the surgery and all treatment modalities are exhausted. In that case, the patient is offered a permanent removal of the stoma, which has a lifelong impact on the patient.

According to the available data, it is possible to prevent the occurrence of LARS through postoperative pelvic floor exercises, however, relevant studies are missing The pelvic floor is a ligament-muscle system that provides dynamic support for the organ systems located in the small pelvis - the urinary system, the genitals, and the intestinal organs.

Exercise of the pelvic floor muscles plays an important role in patients suffering from incontinence, pelvic organ prolapse, or rectal prolapse. Strengthening the muscles can serve as a follow-up treatment after surgical procedures including prevention of LARS.

The resulting knowledge of the possibility of preventing LARS will have a fundamental impact on clinical practice and patient management.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive functions make it possible to understand and sign the patient's informed consent and consent to participate in the study
* Surgical procedure - mini-invasive low anterior rectal resection

Exclusion Criteria:

* not agreeing to participate in the study
* request to practice pelvic floor exercises despite being in the control group
* non-compliance
* serious psychiatric diagnoses

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The number of participants who develop (or what degree) LAR syndrome with or without pelvic floor exercises after LAR, ascertained by LARS questionnaire. | 4 weeks
  Patients may develop varying degrees of functional impairment - defecation urgency, fecal incontinence, increased frequency of stool, fragmentation and numerous bowel movements in a short period, problems with emptying or incomplete stool evacuation, increased intestinal flatulence, diarrhea, constipation or change in stool consistency. Participants will exercise at home. 1,6,12 months after surgery, the Low Anterior Resection Syndrome (LARS) questionnaire will be sent to patients. LARS questionnaire contains 5 questions about bowel functions. It is officially translated into the Slovak language. Final score range between 0-42. 0-20: NO LARS, 21-29: minor LARS, 30 - 42: major LARS.

SECONDARY OUTCOMES:
Adherence of patients to prescribed home exercise after surgery, determined by the Exercise Adherence Rating Scale (EARS) | 4 weeks
  The results can be significantly limited by the patient's actual exercise at home. One month after surgery a 16-item EARS questionnaire using a 5-point Likert scale will be sent to patients. 0 = completely agree to 4 = completely disagree. Summed score range from 0 to 64. Positively phrased items are reversed scored so that a higher overall adherence score indicates better adherence to exercise.

OTHER OUTCOMES:
Quality of life after LAR measured by WHOQOL - BREF | 1 - 12 months after LAR
  Low anterior resection syndrome is a significant factor reducing the quality of life. 1,6,12 months after surgery the WHO Quality of Life Questionnaire - BREF will be sent to patients. It is a 0-100 scale. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Ľubomír Marko, MD,ass. prof, Study Director — F. D. Roosevelt University Hospital; Barbara Mrázová, MD,MPH, Study Chair — F. D. Roosevelt University Hospital
Locations (1):
- F.D.Roosevelt University Hospital in Banská Bystrica, Banská Bystrica, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Demographics, diagnosis, TNM stage, histology, complications, questionaires
Time Frame: 5th June 2024 for at least 5 years
Access Criteria: EU Open Research Repository
URL: https://zenodo.org/records/11486092

REFERENCES:
- [Background] Allgayer H, Dietrich CF, Rohde W, Koch GF, Tuschhoff T. Prospective comparison of short- and long-term effects of pelvic floor exercise/biofeedback training in patients with fecal incontinence after surgery plus irradiation versus surgery alone for colorectal cancer: clinical, functional and endoscopic/endosonographic findings. Scand J Gastroenterol. 2005 Oct;40(10):1168-75. doi: 10.1080/00365520510023477. PMID 16165701
- [Background] Asnong A, D'Hoore A, Van Kampen M, Wolthuis A, Van Molhem Y, Van Geluwe B, Devoogdt N, De Groef A, Guler Caamano Fajardo I, Geraerts I. The Role of Pelvic Floor Muscle Training on Low Anterior Resection Syndrome: A Multicenter Randomized Controlled Trial. Ann Surg. 2022 Nov 1;276(5):761-768. doi: 10.1097/SLA.0000000000005632. Epub 2022 Jul 27. PMID 35894434
- [Background] Laforest A, Bretagnol F, Mouazan AS, Maggiori L, Ferron M, Panis Y. Functional disorders after rectal cancer resection: does a rehabilitation programme improve anal continence and quality of life? Colorectal Dis. 2012 Oct;14(10):1231-7. doi: 10.1111/j.1463-1318.2012.02956.x. PMID 22268662
- [Background] Liu CH, Chen CH, Lee JC. Rehabilitation exercise on the quality of life in anal sphincter-preserving surgery. Hepatogastroenterology. 2011 Sep-Oct;58(110-111):1461-5. doi: 10.5754/hge11160. Epub 2011 Jul 15. PMID 21940307
- [Background] Lin KY, Granger CL, Denehy L, Frawley HC. Pelvic floor muscle training for bowel dysfunction following colorectal cancer surgery: A systematic review. Neurourol Urodyn. 2015 Nov;34(8):703-12. doi: 10.1002/nau.22654. Epub 2014 Aug 23. PMID 25156929
- [Background] Pucciani F, Ringressi MN, Redditi S, Masi A, Giani I. Rehabilitation of fecal incontinence after sphincter-saving surgery for rectal cancer: encouraging results. Dis Colon Rectum. 2008 Oct;51(10):1552-8. doi: 10.1007/s10350-008-9312-6. Epub 2008 May 2. PMID 18452041
- [Background] Emile SH, Garoufalia Z, Barsom S, Horesh N, Gefen R, Zhou P, Wexner SD. Systematic review and meta-analysis of randomized clinical trials on the treatment of low anterior resection syndrome. Surgery. 2023 Jun;173(6):1352-1358. doi: 10.1016/j.surg.2023.02.010. Epub 2023 Apr 1. PMID 37012144